CLINICAL TRIAL: NCT07042841
Title: the Study on AI-Integrated Fully Quantitative Treatment Decision and Surgical Planning System for Liver Cancer
Brief Title: AI-Driven Quantitative Decision and Surgical Planning System for Liver Cancer
Status: Enrolling by invitation | Type: Observational
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Principal Investigator, Shuo Jin, Associate Chief Physician, Beijing Tsinghua Chang Gung Hospital
Other Study IDs: 25293-0-01
Record Dates: First submitted 2025-06-18; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Liver Cancer, Adult
Keywords: Liver Cancer; Artificial Intelligence; Computer-Aided Diagnosis; Multimodal Image Fusion; Pathology-CT Registration
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HCC Positive Group: HCC-positive with liver lesion
- HCC Negative Lesion Group: HCC-negative with liver lesion
- Non-Lesion Control Group: No liver lesion

SUMMARY:
This study aims to develop and validate an integrated AI-powered system for liver cancer that includes intelligent tumor boundary detection, micro-metastasis prediction, staging, treatment decision-making, and surgical planning. The system builds upon prior 3D reconstructions of liver, vessels, and bile ducts. In a retrospective multi-center, self-controlled, fully crossed multi-reader multi-case clinical trial, the researchers will compare diagnostic accuracy, staging, and planning performance between AI-assisted reads and conventional reads using CT images and pathological gold standards.

DETAILED DESCRIPTION:
Background Precise tumor boundary definition on preoperative imaging is often unreliable, and regional disparities in healthcare resources limit personalized decision-making. Currently, no comprehensive AI system integrates imaging, pathology, staging, decision, and surgical planning for liver cancer.

Objectives 1: Develop a pathological-tumor-boundary evaluation system based on whole-slide pathology and CT registration. 2: Build models to predict tumor boundary and satellite micro-metastasis from CT images using deep learning and radiomics. 3: Integrate staging modules (Child-Pugh, ECOG-PS, CNLC/BCLC) and generate individualized treatment recommendations. 4: Create a surgical planning platform that calculates liver remnant volume, vascular invasion metrics, anatomical variants, and performs virtual resections. 5: Validate the system in a retrospective self-controlled multi-reader multi-case study across multiple centers.

Methods Tumor boundary & micro-metastasis prediction: Register 3D whole-slide pathology of resected specimens to preoperative CT using multiplanar reconstruction; pathologists annotate tumor and satellite lesions; train deep-learning models to predict pathological boundaries and micro-metastasis regions. Validate in 100 cases with pathological CT comparison. Decision modules: Automatically compute Child-Pugh and ECOG-PS scores from labs and records; integrate with tumor metrics and PV invasion to achieve CNLC/BCLC staging and generate decision suggestions. Surgical planning: Calculate functional liver volume requirements per consensus, estimate standard liver volume (SLV), tumor-bearing segment volume, future liver remnant (FLR/SLV), flag unsafe resections; analyze vascular invasion level, length, and perfusion territory; detect portal/bile anatomical variants for injury warnings; perform virtual anatomical and non-anatomical resections with margin control and risk predictions. Clinical validation: Conduct a retrospective, fully-crossed multi-reader multi-case trial: randomized CT reading by surgeons/radiologists with and without software assistance, separated by washout periods. Evaluate primary endpoints: AFROC-AUC for lesion detection, LROC-AUC for HCC diagnosis. Secondary endpoints include sensitivity, specificity, ROC-AUC, diagnostic consistency (Kappa), size/count accuracy (<5% error), staging concordance, and reading time.

Study population Adult participants with dynamic contrast-enhanced liver CT, including HCC-positive, HCC-negative lesion-positive, and lesion-negative cases. Exclude cases with incomplete liver imaging, heavy noise, prior liver resection, or unreadable CT.

Statistical analysis Compare AUCs between AI-assisted and manual reading; non-inferiority established if lower bound of 95% CI > 0. Secondary metrics include sensitivity, specificity, consistency, reading time, and staging accuracy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Dynamic contrast-enhanced CT scan of the liver is available. 2. Age ≥ 18 years. 3. CT image slice thickness ≤ 5 mm. 4. An official CT report is available. 5. Meets at least one of the following subcategories:HCC-positive with liver lesion: CT report suggests suspected hepatocellular carcinoma (HCC), and complete hospitalization records are available to assess CNLC staging (including performance status, Child-Pugh classification, and extrahepatic metastasis). HCC-negative with liver lesion: CT report indicates at least one liver-occupying lesion, but not suspected to be HCC. No liver lesion: CT report indicates no liver-occupying lesion.

Exclusion Criteria:

* 1. Incomplete liver coverage in CT images. 2. Severe noise artifacts in CT images. 3. History of liver resection or significant anatomical/volume alterations of the liver. 4. Deemed unsuitable for inclusion by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study aims to include adult patients (≥18 years old) who have undergone dynamic contrast-enhanced CT imaging of the liver. The population will consist of three groups:
  HCC-positive group (Group 1): Patients with liver lesions diagnosed as suspected hepatocellular carcinoma (HCC) based on CT imaging reports, and with complete clinical records for assessment of CNLC staging, Child-Pugh score, and extrahepatic metastasis.
  HCC-negative with liver lesion group (Group 2): Patients with liver lesions identified on CT imaging but without HCC diagnosis, and without clear evidence of extrahepatic metastasis.
  Non-lesion control group (Group 3): Patients with no liver lesions identified on CT imaging, serving as the control group.
  All participants will have a CT imaging slice thickness of ≤5 mm, and must be capable of providing complete imaging reports and medical records. The study will target approximately 300 participants across these groups.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-06-30 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of the intelligent liver cancer diagnosis and surgical planning system | At the time of surgery.
  The diagnostic accuracy will be evaluated by comparing the system's prediction of tumor boundaries and microvascular invasion with pathological gold standards.

CONTACTS AND LOCATIONS:
Overall Officials: Shuo Jin, PhD, Principal Investigator — Beijing Tsinghua Chang Gung Hospital
Locations (1):
- Beijing Tsinghua Chang Gung Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No